CLINICAL TRIAL: NCT05915156
Title: Transition in Care From Post-acute Services for the Elderly in Quebec: A Pilot Impact Evaluation Study
Brief Title: Transition in Care From Post-acute Services for the Elderly in Quebec
Acronym: PAHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal (Other)
Collaborators: McGill University (Other); Université du Québec à Trois-Rivières (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Diana Zidarov, Principal investigator, Centre for Interdisciplinary Research in Rehabilitation of Greater Montreal
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CIUSSS-SMHC-20-21
Record Dates: First submitted 2023-05-31; First posted 2023-06-22 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Older Adults; Rehabilitation; Physical Therapy; Functional Independence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-acute home physiotherapy program (PAHP) (Other): This health services research aimed to assess the effects of a post-acute home physiotherapy program that was designed to provide home physiotherapy services to patients recently discharged from acute or post-acute care.
  Interventions: Other: Post-acute home physiotherapy program

INTERVENTIONS:
Other: Post-acute home physiotherapy program — This health services research assessed the effects of a post-acute home physiotherapy program that was designed to provide physical rehabilitation services to older adults recently discharged from acute or post-acute care. Under this program, every patient was attended by a physiotherapy technologist within 48 hours of being discharged and received home physiotherapy for a minimum of three days per week for a maximum of eight weeks.

SUMMARY:
An early discharge of frail elderly individuals from post-acute care services may lead to a decline in their ability to perform daily activities and cause social, emotional, and psychological distress. Montreal West Island Integrated University Health and Social Services Center in Quebec implemented a pilot program called Post-Acute Home Physiotherapy (PAHP) to address this concern. This program aimed to provide a timely and intense out-patient physiotherapy service to ensure maintenance and optimization of the physical capacities acquired in post-acute care and also to contribute acceleration of the turnover of rehabilitation beds. The objective of this study was to assess the impact of the PAHP program on the functional independence, physical and mental health of elderly individuals, as well as their safety. Additionally, it aimed to identify the healthcare needs, both physical and psychological, of elderly individuals after their discharge from post-acute care services.

DETAILED DESCRIPTION:
Seniors play a key role in our society by participating in social activities, volunteering, and for some, working past the age of 80. By 2030, one out of 4 Canadians will be over the age of 65 and life expectancy will raise to 86.2 years for women and 82.9 for men. The global share of older people will continue to grow as a proportion of the world population, reaching 21.1% by 2050. While people are living longer almost everywhere, including in Canada, the prevalence of disabilities and multimorbidity is increasing as the population ages. Multimorbidity, which is defined as the coexistence of two or more chronic conditions, becomes the norm. In Canada, the overall prevalence of multimorbidity for people aged 40 years and over was 26.5% in 2011/12 and this prevalence increases substantially to 66.3 % for people aged ≥ 85 years. This brings a tremendous challenge to the Canadian healthcare system where high healthcare users, representing only 0.5% of the population aged 50 to 74 and 2.6% of those aged 75 or older, but accounting for about half of all hospital days (45.6% and 56.1%, respectively) recorded for people of these ages.

Hospitalization and prolonged stays in acute care can lead to a functional decline which is one of the most common negative outcomes of hospitalization. Post-hospitalization functional decline has been shown to be sustained up to one year following discharge, and non-recovery to baseline functional status has been associated with increased risk of re-hospitalization, prolonged disability, and death (up to three years). This loss of functional capacity in the elderly raises the need for more innovative and specialized care to help restore and promote seniors' independency after stays in acute care settings. Post-acute care is a set of services and an approach to manage and restore human activity. Post-acute care includes all services needed by end-users requiring rehabilitation to regain functional autonomy. Instead of being discharged from acute care back home or directly to nursing homes, many seniors first transition to post-acute care to receive specialized inpatient and/or outpatient rehabilitation.

In order to provide a timely and intense out-patient physiotherapy service to ensure maintenance and optimization of the physical capacities acquired in post-acute care and also to contribute acceleration of the turnover of rehabilitation beds, the MWI IUHSSC then created a pilot program in November 2017, the Post-acute home physiotherapy program or PAHP. The PAHP program was built in accordance to INESSS recommendation to address the rehabilitation needs of clients ready to return home after transiting in a post-acute facility, but still requiring rehabilitation to maximize their autonomy.

The PAHP program was implemented across the 4 local care centres of the MWIIUHSSC's territory between May 2018-May 2019 serving 163 clients. PAHP was designed for all elderlies in need for additional rehabilitation to be seen by a physical therapist technologist within 48hrs of being discharged from post-acute care and receive physical therapy 3 days/week for a period of 6 weeks. However, the impact of the PAHP program and whether it addresses the healthcare needs of the older people is unknown.

The main objective of this study is to assess the effects of the pilot PAHP program on various aspects of an individual's well-being. These aspects include functional independence, physical and mental health, and overall safety. Additionally, the study aims to identify the physical, mental, and psychological needs of elderly individuals after they have been discharged from post-acute services.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥60 years
* Discharged home with/without home care services
* French or English fluency

Exclusion Criteria:

- Patients were excluded if they had an unstable medical, psychiatric, and post-surgical condition or a severe cognitive impairment (based on the assessment of the rehabilitation team).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Functional Independence Measure | Change from week start of PAHP program (week 0) to end of program (week 8), 3-month follow-up (week 20)
  Change in the Functional Independence Measure between 3 assessment points: week 0, week 8 and week 20. The FIM assesses an individual's independent performance in various areas, including self-care, sphincter control, transfers, locomotion, communication, and social cognition. This assessment consists of 18 items, and each item is assigned a score ranging from 1 to 7. The total score ranges from 18 (indicating the lowest level of independence and requiring significant assistance) to 126 (reflecting a high level of independence and minimal assistance needed).

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System Global-10 survey | Change from week start of PAHP program (week 0) to end of program (week 8), 3-month follow-up (week 20)
  Change in the Patient-Reported Outcomes Measurement Information System Global-10 between 3 assessment points: week 0, week 8 and week 20. The PROMIS Global 10 will be used to assess self-reported perception of health, physical, mental and social health, as well quality of life with a Likert scale of 5 points.
Patient Global Impression of Change Scale | Discharge from PAHP program (Week 8)
  The Patient Global Impression of Change Scale will be used to assess participants' perception of their level of improvement or deterioration of their physical function at discharge from the PAHP program (week 8). An 11-point Likert scale will be used with options ranging from "very much worse" to "completely recovered".
Evaluation of safety parameters (Fall incidence, emergency visits, re-hospitalizations) | Discharge from PAHP program (week 8) and at 3-month follow-up (week 20)
  Change in safety parameters will be assessed between discharge (week 8) from the program and at follow-up (week 20). The self-report of elderly individuals regarding the number of fall incidence, emergency visits, re-hospitalizations with respect to their principal diagnosis were recorded.
Camberwell Assessment for the Need of the Elderly questionnaire | Admission at PAHP program (week 0) and discharge from the program (week 8)
  Change in the Camberwell Assessment for the Need of the Elderly questionnaire will be assessed between admission (week 0) and discharge from the program (week 8). This questionnaire is used to assess the met and unmet physical, psychological, social and environmental care needs (24 domains) from the perspective of the elderly individual. In this questionnaire, for each domain, there is a question about a particular need. Responses are rated on a three-point scale where 0 means no need, 1 - met need (problem receiving proper intervention) and 2 - unmet need (problem left without optimal intervention).

CONTACTS AND LOCATIONS:
Overall Officials: Diana Zidarov, PhD, Principal Investigator — Centre de Recherche Interdisciplinaire en Réadaptation
Locations (6):
- Canada (6):
  - CLSC de Dorval-Lachine, Lachine, Quebec
  - CLSC de LaSalle, LaSalle, Quebec
  - LaSalle Hospital, LaSalle, Quebec
  - CLSC de Pierrefonds, Pierrefonds, Quebec
  - CLSC du Lac-Saint-Louis, Pointe-Claire, Quebec
  - Ste. Anne's Hospital, Sainte-Anne-de-Bellevue, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghai S, Chasse K, Renaud MJ, Guicherd-Callin L, Bussieres A, Zidarov D. Transition of care from post-acute services for the older adults in Quebec: a pilot impact evaluation. BMC Health Serv Res. 2024 Apr 3;24(1):421. doi: 10.1186/s12913-024-10818-2. PMID 38570840